CLINICAL TRIAL: NCT01072981
Title: A Phase III Study of Chemotherapy and Chemoradiotherapy With or Without Algenpantucel-L (HyperAcute®-Pancreas) Immunotherapy in Subjects With Surgically Resected Pancreatic Cancer
Brief Title: Immunotherapy Study for Surgically Resected Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLG0405; OBA# 0912-1013 (Other: Office of Biotechnology Activities)
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Vaccine Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Algenpantucel-L; Gemcitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HyperAcute-Pancreas Immunotherapy + Standard of Care (Experimental): *Adjuvant Standard of Care Treatment (SOC) consisting of gemcitabine with or without 5FU chemoradiation + HyperAcute Immunotherapy
  Interventions: Biological: HyperAcute-Pancreas Immunotherapy; Drug: Gemcitabine; Radiation: 5FU Chemoradiation
- Standard of Care alone (Active Comparator): *Adjuvant Standard of Care Treatment (SOC) consisting of gemcitabine with or without 5FU chemoradiation Alone
  Interventions: Drug: Gemcitabine; Radiation: 5FU Chemoradiation

INTERVENTIONS:
Biological: HyperAcute-Pancreas Immunotherapy — Up to 18 immunizations of 300 million immunotherapy cells
  Other Names: HAPa-1 and HAPa-2 immunotherapy components
  Arms: HyperAcute-Pancreas Immunotherapy + Standard of Care
Drug: Gemcitabine — Gemcitabine 1000 mg/m2/day once a week for 3 weeks
  Other Names: Gemzar
Radiation: 5FU Chemoradiation — 5FU 200-250 mg/m2/day over 5 1/2 weeks with radiation.
  Other Names: Fluorouracil

SUMMARY:
The purpose of this study is to assess overall survival after treatment with a regimen of adjuvant therapy (Gemcitabine alone or with 5-FU chemoradiation) with or without HyperAcute®-Pancreas (algenpantucel-L) immunotherapy in subjects who have undergone surgical resection.

DETAILED DESCRIPTION:
Unfortunately, despite the best clinical efforts and breakthroughs in biotechnology, most patients diagnosed with pancreatic cancer continue to die from the rapid progression of their disease. The primary reason for this is that the disease is typically without symptoms until significant local and/or distant spread has occurred and is often beyond the chance for cure at the time of the diagnosis. The lack of any treatment to significantly increase long term survival rates is reflected by the poor outcomes associated with this disease, specifically time to disease progression and overall survival.

These disappointing facts typically shape discussions of treatment options for patients with this disease. However, another important part of the body is now being looked at as a target for therapy against this disease -- the immune system. Scientists have clearly shown that pancreatic tumor cells produce a number of defective proteins, or express normal proteins in highly uncharacteristic ways, as part of this cancer. In some cancers, these abnormalities can cause an immune response to the cancer cells much in the way one responds to infected tissue. In progressive cancers however, the immune system fails to identify or respond to these abnormalities and the cancer cells are not attacked or destroyed for reasons not yet fully understood. This clinical trial proposes a new way to stimulate the immune system to recognize the abnormal components found in pancreatic cancer cells and to stimulate an immune response that destroys or blocks the growth of the cancer.

This new method of treatment helps the immune system of pancreatic cancer patients to "identify" the cancerous tissue so that it can be eliminated from the body. As an example, most people are aware that patients with certain diseases may require an organ transplant to replace a damaged kidney or heart. After receiving their transplant these patients receive special drugs because they are at great danger of having an immune response that destroys or "rejects" the transplanted organ. This "rejection" occurs when their immune system responds to differences between the cells of the transplanted organ and their own immune system by attacking the foreign tissue in the same way as it would attack infected tissue. When the differences between foreign tissues and the patient's body are even larger, perhaps like differences between organs from pigs and the immune system cells of humans, the rejection is very rapid, highly destructive and the immunity it generates is long lasting. This is called hyperacute rejection and the medicine used to immunize patients in this protocol tries to harness this response to teach a patient's immune system to fight their pancreatic cancer just as the body would learn to reject a transplanted organ from an animal.

To do this, the investigators have placed a mouse gene into human pancreatic cancer cells so that the immune system will easily recognize them as foreign, stimulating the patient immune system to attack the vaccine cells just as they would any other animal cells. As part of the process of destroying the immunotherapy cells, the patient immune system is stimulated to identify as many differences from normal human as possible. This extra stimulation is thought to encourage immune responses against the pancreatic cancer in the patient based on shared abnormalities of pancreatic cancer vaccine cells and the patient's pancreatic cancer cells.

In this experimental therapy, patients are given injections of an immunotherapy consisting of two types of cancer cells that the investigators have modified to make them more easily recognized and attacked by the immune system. The investigators propose to test this new treatment in patients with pancreatic cancer who have undergone tumor removal surgery but remain at extremely high risk of disease progression to demonstrate that treatment with the immunotherapy increases the time until the tumor recurs or increases overall survival when given in combination with the current standard of care therapy for this disease.

For more information, please see our study specific website: www.pancreaticcancer-clinicaltrials.com

ELIGIBILITY:
Inclusion Criteria:

* A histological diagnosis of adenocarcinoma of the pancreas confirmed by pathology.
* American Joint Committee on Cancer (AJCC) Stage I or II Pancreatic carcinoma. Patients must have undergone surgical resection for the tumor and extent of resection must be either R0 (complete resection with grossly and microscopically negative margins of resection) or R1 (grossly negative but positive microscopically margins of resection).
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Serum albumin ≥2.0 gm/dL.
* Expected survival ≥6 months.
* Subjects must be able to take in adequate daily calorie intake based on judgment of clinical investigator.
* Adequate organ function including:
* A. Marrow: white blood cells (WBC) ≥3000/mm3 and platelets ≥100,000/mm3.
* B. Hepatic: serum total bilirubin ≤2 x ULN mg/dL, ALT (SGPT) and AST (SGOT) ≤3 x upper limit of normal (ULN).
* C. Renal: serum creatinine (sCr) ≤2.0 x ULN, or creatinine clearance (Ccr) ≥30 mL/min.
* First vaccination must be within 10 weeks after surgery.
* Patients must have the ability to understand the study, its inherent risks, side effects and potential benefits and be able to give written informed consent to participate. Patients may not be consented by a durable power of attorney (DPA).
* All subjects of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental product, and for one month after the last immunization.

Exclusion Criteria:

* Age <18-years-old.
* Active metastases. Suspicious lesions on CT scans must be reviewed by a second, different reviewer. If active disease not ruled out by second, different reviewer (at clinical institution), a positron emission tomography (PET) CT or further imaging tests or histology may be needed to rule out disease before enrollment is allowed.
* Other malignancy within five years, unless the probability of recurrence of the prior malignancy is <5% as determined by the Principal Investigator based on available information. Patient's curatively treated for squamous and basal cell carcinoma of the skin or patients with a history of malignant tumor in the past that have been disease free for at least five years are also eligible for this study.
* History of organ transplant.
* Current, active immunosuppressive therapy such as cyclosporine, tacrolimus, etc.
* Subjects taking chronic systemic corticosteroid therapy for any reason are not eligible. Subjects may receive steroids as prophylactic anti-emetics, not to exceed 10 mg Decadron weekly. Subjects may also receive pulse doses for Gemcitabine hypersensitivity, not to exceed Decadron 8 mg twice a day (BID) x 3 days prior to start day of Gemcitabine. Subjects receiving inhaled or topical corticosteroids are eligible. Subjects who require chronic systemic corticosteroids after beginning vaccination, will be removed from study.
* Significant or uncontrolled congestive heart failure (CHF),myocardial infarction or significant ventricular arrhythmias within the last six months.
* Active infection or antibiotics within 48 hours prior to study,including unexplained fever (temp > 38.1C).
* Autoimmune disease (e.g., systemic lupus erythematosis (SLE), rheumatoid arthritis (RA), etc.). Patients with a remote history of asthma or mild active asthma are eligible.
* Other serious medical conditions that may be expected to limit life expectancy to less than 2 years (e.g., liver cirrhosis) or a serious illness in medical opinion of the clinical investigator.
* Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc.).
* A known allergy to any component of the HyperAcute® immunotherapy.
* Pregnant or nursing women due to the unknown effects of vaccination on the developing fetus or newborn infant. (For patients with child bearing potential, a βHCG must be completed within 14 days of first vaccination).
* Known HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2010-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess overall survival | Approximately 41 months and 48 months

SECONDARY OUTCOMES:
The secondary objective is to assess disease free survival and to conduct correlative scientific studies of subject samples to determine the mechanism of any observed anti-tumor effect. | Approximately 41 months and 48 months

CONTACTS AND LOCATIONS:
Locations (75):
- United States (75):
  - University of Alabama, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Sutter Institute for Medical Research, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Stamford Hospital, Stamford, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Boca Raton Hospital, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - University of Miami, Miami, Florida
  - USF Tampa General, Tampa, Florida
  - MOFFITT, Tampa, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Northwestern University, Chicago, Illinois
  - Northshore University Health Systems, Evanston, Illinois
  - Edward H. Kaplan, MD and Associates, Skokie, Illinois
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University, Indianapolis, Indiana
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico, Albuquerque, New Mexico
  - Mount Sinai Medical Center, New York, New York
  - Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health Comprehensive Cancer Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Western, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Greenville Health System, Greenville, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Texas Health Sciences, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Lynchburg Hematology-Oncology Clinic, Inc., Lynchburg, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington- Seattle Cancer Center Alliance, Seattle, Washington
  - Vince Lombardi Cancer Clinic, Green Bay, Wisconsin
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Hardacre JM, Mulcahy M, Small W, Talamonti M, Obel J, Krishnamurthi S, Rocha-Lima CS, Safran H, Lenz HJ, Chiorean EG. Addition of algenpantucel-L immunotherapy to standard adjuvant therapy for pancreatic cancer: a phase 2 study. J Gastrointest Surg. 2013 Jan;17(1):94-100; discussion p. 100-1. doi: 10.1007/s11605-012-2064-6. Epub 2012 Nov 15. PMID 23229886